CLINICAL TRIAL: NCT06049186
Title: Comparison of Live Birth Rates Between Calorie-restricted Diets and Metformin Interventions Prior to Ovulation Induction Therapy in Patients With Overweight/Obese Polycystic Ovary Syndrome Combined With Infertility
Brief Title: CRD vs. Met in Patients With Obese PCOS Infertility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: RenJi Hospital (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD vs. Met in PCOS
Record Dates: First submitted 2023-08-31; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Caloric Restriction; Metformin

STUDY DESIGN:
Intervention Model Description: Comparison of live birth rates between calorie-restricted diets and metformin interventions prior to ovulation induction therapy in patients with overweight/obese polycystic ovary syndrome combined with Infertility.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRD group (Experimental): Patients in the calorie-restricted diet (CRD) group will have strict calorie-restriction diets for 8 weeks and then weight stability for 4 weeks.
  Interventions: Behavioral: CRD
- Control group (Active Comparator): Patients in the control group will receive regular diets and metformin 1500 mg daily for 12 weeks. Participants allocated to the control group are followed by the conventional approach (usual care) based on regular visits respecting the usual schedule dictated by the rules of general practice.
  Interventions: Drug: Metformin

INTERVENTIONS:
Behavioral: CRD — During the initial 8 weeks of the trial, polycystic ovary syndrome (PCOS) patients are instructed to follow a diet of 1200 to 1500 kcal per day supervised by dietitians. The CRD includes a combination of 40 to 55% of calories from carbohydrates, 15 to 20% from protein, and 20 to 30% from fat; this regimen represented approximately 75% of the participants' daily caloric intake at baseline. All the participants receive dietary counseling daily during the trial.
  Other Names: Calorie-restricted diet
  Arms: CRD group
Drug: Metformin — After randomization, patients entering the metformin group will be given 1500 mg daily (bid/tid) metformin and regular diets as control. Participants allocated to the control group are followed by the conventional approach (usual care) based on regular visits respecting the usual schedule dictated by the rules of general practice.
  Other Names: Metformin treatment
  Arms: Control group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common gynecological endocrine disease and a major cause of anovulatory infertility in reproductive-aged women. From 2010 to 2020, it was found that the prevalence of PCOS in reproductive-aged women in China reached 7.8%, an increase of 65% over 10 years ago. Many of them are overweight or obese. Weight loss including diet modifications can significantly reduce reproductive and metabolic disorders of PCOS and is recommended as a first step in the treatment of overweight or obese women with PCOS. Many weight loss programs have been proposed, including calorie-restriction diet (CRD) intervention. Whether CRD intervention prior to ovulation induction therapy could improve live birth rates in overweight/obese PCOS women has not been illustrated.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a common gynecological endocrine disease and a major cause of anovulatory infertility in reproductive-aged women. Rotterdam criteria state the definition of PCOS is that women must present with two of the following three signs/symptoms-hyperandrogenism, chronic anovulation/oligomenorrhea, and polycystic ovaries-in the absence of other diseases that promote these symptoms. From 2010 to 2020, it was found that the prevalence of PCOS in reproductive-aged women in China reached 7.8%, an increase of 65% over 10 years ago. Many of them are overweight or obese. Weight loss including diet modifications can significantly reduce reproductive and metabolic disorders of PCOS and is recommended as a first step in the treatment of overweight or obese women with PCOS. Many weight loss programs have been proposed, including calorie-restriction diet (CRD) intervention. Whether CRD intervention prior to ovulation induction therapy could improve live birth rates in overweight/obese PCOS women has not been illustrated. This research is aimed to evaluate whether CRD intervention prior to ovulation induction could promote reproductive health in overweight or obese PCOS women with fertility requirements and provide an evidence-based nutrition advice for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of polycystic ovary syndrome (PCOS) based on the Rotterdam diagnostic criteria;
2. age 20-35 years old;
3. a body-mass index over 23;
4. have requirements for fertility.

Exclusion Criteria:

1. acute or chronic viral hepatitis;
2. serious liver dysfunction or chronic kidney disease;
3. serious cardiovascular or cerebrovascular disease;
4. patients with a history of acute/chronic infection, severe cardiovascular and cerebrovascular diseases, and malignant tumors;
5. have drugs for PCOS such as glucocorticoids and anti-androgen drugs (spironolactone, cyproterone acetate, flutamide, etc.) within 3 months;
6. congenital or secondary uterine abnormalities;
7. use of medications that affect weight or energy balance such as Metformin within 3 months;
8. undergoing weight loss treatment (weight change greater than 5% in the past 3 months) or have a history of gastrointestinal surgery;
9. tubal obstruction;
10. the total number of motile sperm of male partner is less than 10 million;
11. any other situations that might affect the trial.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 406 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Live birth during the period of ovulation induction | 18 months
  Live birth will be defined as the delivery of one or more living infants (≥22 week's gestation or birth weight more than 500g). The outcome could be assessed by clinical data and clinical diagnosis.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) | Baseline period and 3 months
  A laboratory test that determines the level of glucose in the blood after an overnight fast, used especially to diagnose diabetes and prediabetes. The normal interval is 3.9-6.1mmol/L. The outcome could be assessed by clinical data and clinical test.
Fasting insulin (FINS) | Baseline period and 3 months
  The level of insulin in the blood during fasting (usually in the morning when fasting). The normal interval is 5~20 μIU. The outcome could be assessed by clinical data and clinical test.
Oral glucose tolerance test (OGTT) | Baseline period and 3 months
  An oral glucose tolerance test (OGTT) is a diagnostic tool used to evaluate how an individual's body metabolizes sugar. Often used to diagnose diabetic conditions, an oral glucose tolerance test requires minimal preparatory measures and may be safely administered during pregnancy. The outcome could be assessed by clinical data and clinical test.
Insulin release test (IRT) | Baseline period and 3 months
  Quantitative oral glucose during fasting increases blood glucose and stimulates pancreatic β cells to release insulin. By measuring plasma insulin levels during fasting and 0.5h, 1h, 2h, and 3h after taking sugar, we can understand the secretion and reserve function of pancreatic β cells, which is also helpful for the classification of diabetes mellitus and guide treatment. The outcome could be assessed by clinical data and clinical test.
Blood lipid | Baseline period and 3 months
  Lipid related indicators include cholesterol, triglycerides. The outcome could be assessed by clinical data and clinical test.
Kidney function index | Baseline period and 3 months
  Blood tests that are included in the kidney function test include measuring for creatinine and blood urea nitrogen (BUN). The outcome could be assessed by clinical data and clinical test.
Liver function index | Baseline period and 3 months
  Liver function index includes alanine aminotransferase (ALT), alkaline phosphatase (ALP) . The outcome could be assessed by clinical data and clinical test.
Free testosterone (FT) | Baseline period and 3 months
  The average serum testosterone concentration is 0.43ng/ml, the high limit is 0.68ng/ml, if more than 0.7ng/m1 (equal to 2.44nmol/L), it is called hypertestosterone, or hyperandrogenemia. The outcome could be assessed by clinical data and clinical test.
Total testosterone (TT) | Baseline period and 3 months
  The normal range of female testosterone is 0.1-0.75ng /ml, testosterone is the main sex hormone of the human body, men and women have secretion, male testosterone secretion is 20-30 times the amount of female testosterone secretion, it is very important to maintain the second sexual characteristics, bone and muscle strength. The outcome could be assessed by clinical data and clinical test.
Sex Hormone Binding Globulin (SHBG) | Baseline period and 3 months
  A globulin synthesized by liver cells that can bind sex hormones, also known as testosterone - estrogen binding globulin or steroidal binding protein, is an important carrier of sex hormones, which can have an important impact on the regulation of sex hormone levels and bioavailability in the body. Clinical detection of SHBG level can provide scientific reference value for disease detection and judgment. The normal interval is 20-130nmol/L for women. The outcome could be assessed by clinical data and clinical test.
Liver transient elastography(TE) | Baseline period and 3 months
  TE may be used to monitor disease progression or regression via serial measurements and to guide further management including treatment. The outcome could be assessed by clinical data and clinical test.
Weight | Baseline period and 3 months
  Unit: kilogram (kg). The outcome could be assessed by clinical data and clinical test.
Height | Baseline period and 3 months
  Unit: meter (m). The outcome could be assessed by clinical data and clinical test.
Body Mass Index (BMI) | Baseline period and 3 months
  BMI = weight (in kg)/ height^2 (in m^2).
Waist circumference | Baseline period and 3 months
  Unit: centimeter (cm). The outcome could be assessed by clinical data and clinical test.
Body fat | Baseline period and 3 months
  Body fat is measured by body fat scale. The outcome could be assessed by clinical data and clinical test.
Lean body weight | Baseline period and 3 months
  Lean body weight refers to the total weight of organs, bones, and muscles. The outcome could be assessed by clinical data and clinical test.
Blood pressure (BP) | Baseline period and 3 months
  Blood pressure is a measurement of the force of blood against the arterial walls when the heart pumps. The pressure is measured in millimeters of mercury (mmHg) and is expressed as two numbers. For example, the optimal BP for an adult is 120 over 80, or 120/80. A pressure reading of 120 over 80 or lower is considered healthy. If the systolic number ranges above 120 to 139 or the diastolic number ranges above 80 to 89, a person is considered to have pre-hypertension. Systolic readings from 140 to 159 or diastolic readings from 90 to 99 are classified as stage 1 hypertension. Systolic measurements of 160 or above or diastolic measurements of 100 or above indicate the severe condition of stage 2 hypertension. The outcome could be assessed by clinical data and clinical test.
Hospital Anxiety and Depression Scale (HADS) | Baseline period and 3 months
  The purpose of the HADS was to screen for clinically significant anxiety and depressive symptoms in medically ill patients. Content The HADS-A includes specific items that assess generalized anxiety including tension, worry, fear, panic, difficulties in relaxing, and restlessness. The total score for the HADS-A can range from 0 to 21. The following guidelines are recommended for the interpretation of scores: 0-7 for normal or no anxiety, 8-10 for mild anxiety, 11-14 for moderate anxiety, and 12-21 for severe anxiety.
Biochemical pregnancy | 8 months
  A pregnancy diagnosed only by the detection of beta hCG in serum or urine. The outcome could be assessed by clinical data and clinical diagnosis.
Ectopic pregnancy | 8 months
  Ectopic pregnancy (EP) is defined as the implantation and development of a fertilized ovum anywhere outside of the uterine cavity. The outcome could be assessed by clinical data and clinical diagnosis.
Pregnancy failure | 8 months
  Pregnancy failure, otherwise termed as pregnancy loss or miscarriage, can occur at different stages during this process and many different pathophysiological mechanisms may be implicated. The outcome could be assessed by clinical data and clinical diagnosis.
Birth weight | 18 months
  Macrosomia is defined in a newborn as a birth weight more than two standard deviations above the mean percentile for gestational age, >90th percentile weight for gestational age, or a birth weight greater than 4000g at term. The outcome could be assessed by clinical data and clinical diagnosis.
Neonatal complications | 18 months
  Neonatal complications include intraventricular hemorrhage, necrotizing enterocolitis, respiratory distress syndrome, bronchopulmonary dysplasia, jaundice. The outcome could be assessed by clinical data and clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Miaoxin Chen, Dr, Study Chair — Shanghai First Maternity and Infant Hospital
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang R, Li Q, Zhou Z, Qian W, Zhang J, Wu Z, Jin L, Wu X, Zhang C, Zheng B, Tan J, Hao G, Li S, Tian T, Hao Y, Zheng D, Wang Y, Norman RJ, Li R, Liu P, Qiao J. Changes in the prevalence of polycystic ovary syndrome in China over the past decade. Lancet Reg Health West Pac. 2022 May 31;25:100494. doi: 10.1016/j.lanwpc.2022.100494. eCollection 2022 Aug. PMID 35669932
- [Background] Lie Fong S, Douma A, Verhaeghe J. Implementing the international evidence-based guideline of assessment and management of polycystic ovary syndrome (PCOS): how to achieve weight loss in overweight and obese women with PCOS? J Gynecol Obstet Hum Reprod. 2021 Jun;50(6):101894. doi: 10.1016/j.jogoh.2020.101894. Epub 2020 Aug 16. PMID 32814159
- [Background] Shahid R, Iahtisham-Ul-Haq, Mahnoor, Awan KA, Iqbal MJ, Munir H, Saeed I. Diet and lifestyle modifications for effective management of polycystic ovarian syndrome (PCOS). J Food Biochem. 2022 Jul;46(7):e14117. doi: 10.1111/jfbc.14117. Epub 2022 Feb 24. PMID 35199348
- [Background] Szczuko M, Kikut J, Szczuko U, Szydlowska I, Nawrocka-Rutkowska J, Zietek M, Verbanac D, Saso L. Nutrition Strategy and Life Style in Polycystic Ovary Syndrome-Narrative Review. Nutrients. 2021 Jul 18;13(7):2452. doi: 10.3390/nu13072452. PMID 34371961
- [Background] Paoli A, Mancin L, Giacona MC, Bianco A, Caprio M. Effects of a ketogenic diet in overweight women with polycystic ovary syndrome. J Transl Med. 2020 Feb 27;18(1):104. doi: 10.1186/s12967-020-02277-0. PMID 32103756